CLINICAL TRIAL: NCT00419679
Title: A Prospective Blinded Study to Evaluate and Characterise an Assay for the Diagnosis of Breast Cancer Using Synchrotron-Derived X-Ray Diffraction of Hair Fibres.
Brief Title: Use of Hair to Diagnose Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fermiscan Ltd (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: FT3.6k-2006
Record Dates: First submitted 2007-01-07; First posted 2007-01-09 (Estimated); Last update posted 2007-01-09 (Estimated); Status verified 2007-01

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; hair; fibre; synchrotron; x-ray diffraction
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Procedure: x-ray diffraction of human hair

SUMMARY:
Study FT3.6k-2006 is a single centre (the Mater Hospital, Sydney), blinded trial of a diagnostic test for breast cancer, with outcomes compared to the gold standard of screening mammogram followed by biopsy where required. This study aims to perform X-ray diffraction analysis of coded hair samples from women with a documented breast health status, to validate the findings of James et al (Nature 398: 33-4, 1999; Int J Cancer 114: 969-72, 2005) who showed that the presence of breast cancer could be detected using synchrotron-derived x-ray diffraction of human hair (scalp or pubic). The aim is also to characterise the sensitivity and specificity of the hair test in detecting breast cancer in a screening setting, and to determine the significance of a positive hair test and a negative mammogram.

DETAILED DESCRIPTION:
The test has the potential to improve the diagnostic (and consequently therapeutic) paradigm for breast cancer.

Women attending a radiology clinic in the Mater Hospital, Sydney, for a mammogram will be invited to participate in the study. A few hairs will be cut from their head or pubic region, put into a coded container and sent to the sponsor for analysis by synchrotron-x-ray diffraction. Although an imperfect standard for a variety of reasons, mammography is the standard screening assay, and confirmation of the pathology of the lesions found by mammography is carried out by biopsy. This will be the standard to which the hair test results will be compared. A negative mammogram will confirm a negative hair test, but a negative mammogram combined with a positive hair diffraction test will need a different approach. In the event of a positive hair test and a negative second read of the mammogram, the patient will be contacted by the referring practitioner. Patients in this category will be offered a breast MRI. A negative breast MRI under these circumstances will be classified as a true negative.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (aged >20) who are undergoing mammography at the Mater Hospital, Sydney, and
* Who are willing and able to provide informed consent; and
* Who have usable scalp and/or pubic hair

Exclusion Criteria:

* Women who have dyed or permed their scalp hair within the previous 6 weeks and whose pubic hair is unavailable;
* Women with a history of breast cancer ever or other cancers (excluding non-melanoma skin cancer and CIN [cervical intra-epithelial neoplasia]) within 5 years.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600
Dates: Start 2006-12

PRIMARY OUTCOMES:
The primary outcome is the determination of the accuracy (sensitivity and specificity) of the x-ray diffraction test for breast cancer using hair. Sensitivity is defined as the proportion of all positive Fermiscan tests that are true positives.

SECONDARY OUTCOMES:
The prevalence of a positive x-ray diffraction hair test and a negative mammogram, and of a negative hair test and a positive mammogram

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Yuile, MBBS (Hons), FRNZCR, Principal Investigator — The Mater Hospital, Sydney
Locations (1):
- The Mater Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Background] James VJ. A place for fiber diffraction in the detection of breast cancer? Cancer Detect Prev. 2006;30(3):233-8. doi: 10.1016/j.cdp.2006.04.001. Epub 2006 Jul 28. PMID 16876335
- [Background] James V, Corino G, Robertson T, Dutton N, Halas D, Boyd A, Bentel J, Papadimitriou J. Early diagnosis of breast cancer by hair diffraction. Int J Cancer. 2005 May 10;114(6):969-72. doi: 10.1002/ijc.20824. PMID 15645416
- [Background] James V. False-positive results in studies of changes in fiber diffraction of hair from patients with breast cancer may not be false. J Natl Cancer Inst. 2003 Jan 15;95(2):170-1. doi: 10.1093/jnci/95.2.170. No abstract available. PMID 12529353
- [Background] Meyer P, James VJ. Experimental confirmation of a distinctive diffraction pattern in hair from women with breast cancer. J Natl Cancer Inst. 2001 Jun 6;93(11):873-5. doi: 10.1093/jnci/93.11.873. No abstract available. PMID 11390537
- [Background] James V, Kearsley J, Irving T, Amemiya Y, Cookson D. Using hair to screen for breast cancer. Nature. 1999 Mar 4;398(6722):33-4. doi: 10.1038/17949. No abstract available. PMID 10078527